CLINICAL TRIAL: NCT04920825
Title: Sacha Inchi Oil Supplementation Among The 3Hs (Hyperglycaemia, Hypertension & Hyperlipidaemia) Patients: A Randomised, Placebo-Controlled, Double-Blinded Human Clinical Trial
Brief Title: Sacha Inchi Oil Supplementation in 3Hs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Dr. Lee Lai Kuan, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: USM/JEPeM/20120710
Record Dates: First submitted 2021-05-26; First posted 2021-06-10 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Endocrine and Metabolic Secondary Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacha Inchi Oil softgel (Active Comparator): Oral Sacha Inchi oil softgel supplement
  Interventions: Dietary Supplement: Sacha Inchi Oil softgel supplement
- Corn oil softgel (Placebo Comparator): Oral corn oil softgel
  Interventions: Dietary Supplement: Corn oil softgel

INTERVENTIONS:
Dietary Supplement: Sacha Inchi Oil softgel supplement — A twice daily supplementation of Sacha Inchi Oil softgel for 12 weeks
  Arms: Sacha Inchi Oil softgel
Dietary Supplement: Corn oil softgel — A twice daily supplementation of Corn Oil softgel for 12 weeks (Placebo)
  Arms: Corn oil softgel

SUMMARY:
The objective of this study is to evaluate the effect of Sacha Inchi Oil supplementation among the 3Hs patients.

DETAILED DESCRIPTION:
Non-communicable diseases (NCDs) are the leading cause of death worldwide. In Malaysia, NCDs account for 67% of premature mortality, and over 70% of disease burden in 2014. In 2016, NCDs were responsible for 71% of the 57 million deaths globally. An estimated 78% of all NCD deaths and 85% of premature adult NCD deaths occurred in low- and middle-income countries. In Malaysia, NCDs contribute to 71% of premature deaths. According to the Malaysian Burden of Disease and Injury Study (2009-2014), cardiovascular and circulatory diseases contributed to 34.8% of deaths. Data from NHMS 2015 showed an increasing trend for diabetes and hypercholesterolaemia but a plateau trend for hypertension. The prevalence of diabetes was from 11.2% (2011) to 13.4% (2015), hypertension from 32.7% (2011) to 30.3% (2015) and hypercholesterolaemia from 35.1% (2011) to 47.7% (2015).

The burden of NCDs has increased substantially over the years. Information from the Global Burden of Disease Study suggests that the biggest contributor amongst the modifiable behavioural risk factors is unhealthy eating. The exposure to an unhealthy diet occurs throughout the lifespan of an individual and accumulates over his/her lifetime. With the increasing prevalence of diabetes and the high prevalence of hypertension and hypercholesterolaemia, it is unlikely that Malaysia will be able to achieve target 3.4 of the United Nations Sustainable Development Goals (of reducing premature mortality due to NCDs). At the current trajectory, it is also unlikely for Malaysia to reach the nine voluntary global targets for the prevention and control of NCDs.

There is an urgent need to reduce exposure to NCD risk factors amongst Malaysians. There are evidences that medical nutrition therapy using nutritional supplements are recommended to treat NCDs. Nutritional supplements contain biologically active ingredients associated with physiological health benefits for preventing and managing chronic diseases, such as hypertension, hyperlipidaemia, and diabetes mellitus . Natural nutraceuticals were a preferable treatment method that has been accepted by consumers and appeared to be generally safe . Among the nutritional supplements used in controlling chronic diseases is the utilisation of long-chain polyunsaturated fatty acids.

Fatty acids (FA) are hydrocarbon chains with a carboxyl group at one end and a methyl group at the other. The carboxyl group is reactive and readily forms ester links with alcohol groups, for example, those on glycerol or cholesterol, in turn, forming acylglycerols (e.g.: triacylglycerols, phospholipids) and cholesterol esters. They have a variable-length carbon chain and can be categorised based on the degree of saturation of their carbon chains. Saturated fatty acids (SFA) possess the maximal number of hydrogen atoms, while monounsaturated fatty acids (MUFA) have one double bond. Fatty acids with double bonds in the hydrocarbon chain are referred to as unsaturated fatty acids; a fatty acid with 2 or more double bonds is called polyunsaturated fatty acids (PUFA). The number of carbon atoms in the chain is denoted by a shorthand nomenclature and the position of the first double bond relative to the methyl (called n) carbon. PUFA can be further subdivided based on the location of the first double bond relative to the methyl terminus of the chain. For example, omega-3 (Ω-3) and omega-6 (Ω-6) FAs are two of the most biologically significant PUFA classes and have their first double bond on either the third or sixth carbon from the chain terminus, respectively . Long-chain Ω-3 and Ω-6 PUFA are synthesised from the essential FAs (EFAs) alpha-linolenic acid (ALA) and linoleic acid (LA), respectively. EFAs cannot be made by the human body and must be obtained through dietary sources. However, animals and humans have the capacity to metabolise EFAs to long-chain derivatives through multiple elongation and desaturation steps.

A high amount of ALA can be found in many nuts . Some Peruvian species that contain this compound in a high percentage is the Sacha Inchi (Plukenetia Volubilis L.). Sacha Inchi is a plant of the Euphorbiaceous family, which grows in the Amazonian forest. The plant, widely cultivated in Peru, has been a component of various native tribal groups of the region. The seeds of Sacha Inchi are of great interest because they contain approximately, on average, 48% oil and 27% proteins. Sacha Inchi seeds have a unique fatty acid composition containing a large amount of unsaturated fatty acids (about 85% polyunsaturation), comprised of approximately 51% linolenic acid (Ω-3) and 34% linoleic acid (Ω-6) . This Peruvian species has been classified as an edible oil with the highest proportion of unsaturated fatty acids7. The oil from Sacha Inchi also contains a high content of gamma- & ∂-tocopherols, it is, despite its high proportion of unsaturated fatty acids, which in turns makes it comparably stable against oxidation. Several in vivo studies have proven that Sacha Inchi can be exquisitely digested. Traditionally, the oil has been used in the preparation of various meals, the seeds are roasted and the leaves are cooked & consumed. SI seeds are also used as a traditional remedy in the Amazon region to treat rheumatic problems and aching muscles . Sacha Inchi oil (SIO) has also been identified as an important source of the healthy Ω-3 and Ω-6 linoleic acyl groups, which are beneficial in controlling cardiometabolic syndrome namely coronary heart disease and hypertension, showing a hypocholesterolaemic effect when used as food supplements.

Literature suggests that Ω-3 and Ω-6 must co-exist or taken in the ratio of 1:1, which is the closest during evolution of humans in order to be beneficial for human health. Common fish oil and nuts have the Ω-3 to Ω-6 variation of 5-13:1 and 1:4-16 respectively. Ω-6 or linoleic acid are not favourable to be ingested in such a tilted ratio as it increases low-density lipoprotein oxidation and severity of coronary atherosclerosis. Clinical studies on high Ω-6/Ω-3 ratio found that when the ratio decreases, the platelet aggregation; the underlying mechanism of atherosclerosis also decreases. A lower Ω-6/Ω-3 ratio also has been found to decrease vascular endothelial growth factor. Too high amount of Ω-6 also inhibits eicosapentaenoic acid incorporation from dietary Ω-3 supplements in human subjects. Throughout a variety of nuts and fishes, Sacha Inchi oil has a 1:1.25 Ω-6 to Ω-3 ratio, approaching the closest of ideal ratio of 1:1. The ideal ratio as demonstrated, could be of relevance to both neurodevelopment and the prevention of neurodegeneration. A target of 1:1 to 2:1 has appeared to be consistent with studies on evolutionary aspects of diet, neurodevelopment, and genetics.

Type 2 Diabetes Mellitus (T2DM), hypertension and hyperlipidaemia are the most common form of NCDs in Malaysia. Prescription of standard and long term medical regimen has long been implemented in managing the illnesses. There is a need to search for some potential complementary medicine to combat 3Hs. The use of Sacha Inchi oil as part of the dietary regimen, or alternative medicine to alleviate the disease progression is the novel research focus among the scientific communities. With the aforementioned, this randomised, placebo-controlled, double-blinded human clinical trial is aimed to determine the efficacy of 12 weeks supplementation of Sacha Inchi oil, a natural blend of polyunsaturated fatty acids among the 3Hs patients. Secondary outcomes include the assessment of vascular implication biomarkers, inflammatory markers, nutritional status, quality of life, mental health, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with 3 simultaneous NCDs (T2DM, hypertension and hyperlipidaemia), for at least 6 months' duration, sub-optimally controlled without clinically manifest complications (retinopathy, diabetic nephropathy, foot ulcer, cardiovascular diseases, chronic kidney disease, aneurysms).
* Male or female
* Pharmacological treated with oral anti-diabetic agents (metformin, sulphonylureas, meglitinides, alpha-glucosidase inhibitors, Thiazolidinediones, Dipeptidyl Peptidase-4 (DPP-4) Inhibitors, or Sodium-glucose Cotransporter 2 (SGLT2) Inhibitors) and/or injecting agents (Glucagon-like Peptide-1 (GLP-1) Receptor Agonists, anti-hypertensive agents (diuretics, beta blockers, calcium channel blockers, ACE inhibitors, angiotensin inhibitor blockers and direct renin inhibitors) and lipid modifying agents (statins, fibrates, PCSK 9 inhibitors, anion exchange resins, niacin and cholesterol absorption inhibitors) as standard medication regimen.
* Chronological age of 18 years and above
* Metabolically stable with baseline biochemical screening taken at least one (1) month before intervention. Values as below:

  * A1c 6.0-8.5%; fasting plasma glucose 6.4-8.5mmol
  * Blood pressure >140/90mmHg - ≤180/110mmHg
  * Total cholesterol (TC) >5.2 mmol/L; high density lipoprotein cholesterol (HDL-C) <1.0 mmol/L (males), <1.2 mmol/L (females); triglycerides (TG) > 1.7 mmol/L, low density lipoprotein cholesterol (LDL-C) >3.4 mmol/L
* Not taking anti-inflammatory supplements (example of the anti-inflammatory supplement: fish oil, flaxseed oil, curcumin extract, ginger extract, spirulina, vitamin C, polyphenol extract blend)

Exclusion Criteria:

* Have been diagnosed with liver diseases (chronic liver failure, cirrhosis, all types of hepatitis), kidney (chronic kidney disease, haemodialysis) or haematological (anaemia, thalassemia, haemophilia) disorders based on pre-screening medical records and during face-to-face interview prior to recruiting. Subjects with identified non-alcoholic steatohepatitis will be excluded through initial AMDI database screening based on liver enzymes blood routine check.
* Active gastric/duodenal ulcer
* Psychiatric disease/mental retardation (bipolar disorder, depression, schizophrenia)
* Cancer (all types), and other diagnosed endocrine disorders apart from type 2 DM such as Cushing's-, Addison's-, Grave's- and Hashimoto's disease, gigantism, acromegaly, hyper- and hypothyroidism.
* Alcohol and drug abuse (self-mentioned or as recorded in the medical card)
* Gestational diabetes mellitus
* Pregnant/lactating. Pregnancy screening test will be conducted for all childbearing age women.
* Hormone replacement therapy (for at least 3 months before entering the study)
* Using herbal remedies (any parts from the plants such as flower, rhizome, seeds, roots, leaves, fruits, stems). Herbal remedies used are medicinal products consisting of a concoction of various plants, used, and believed as disease management and prevention is excluded. Meanwhile ulam (traditional Malay salad) is defined as fresh or raw green salad that can be eaten with fermented sauce, herbs, or spices as side dishes . Ulam consumers will be recruited in the study as ulam is considered as salad consumption.
* Use of steroids, chemotherapy, immunosuppressants or radiotherapy
* Currently under another supplementary program. Other supplementary programmes are defined as a person is enrolled in another clinical trial with the intention-to-treat drugs/supplements. Vitamins or any other supplements (e.g: iron) is included if the outcome is to see to the effect of disease management or prevention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change of Glycated haemoglobin (HbA1c) | Baseline and 12 weeks
  Glycated hemoglobin (HbA1c) is measured in %
Change of Fasting plasma glucose (FPG) | Baseline and 12 weeks
  Fasting plasma glucose (FPG) is measured in mmol/L
Change of fasting serum insulin | Baseline and 12 weeks
  Fasting serum insulin will be measured by radioimmunoassay kit
Change of blood pressure level | Baseline and 12 weeks
  Blood pressure will be recorded as systolic and diastolic, and recorded as mmHg
Change of total cholesterol (TC) | Baseline and 12 weeks
  Total cholesterol (TC) is measured in mmol/L
Change of low density lipoprotein-cholesterol (LDL-C) | Baseline and 12 weeks
  Low density lipoprotein-cholesterol (LDL-C) is measured in mmol/L
Change of high density lipoprotein-cholesterol (HDL-C) | Baseline and 12 weeks
  High density lipoprotein-cholesterol (HDL-C) is measured in mmol/L
Change of triglyceride (TG) | Baseline and 12 weeks
  Triglyceride (TG) is measured in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Lai kuan Lee, PhD, Principal Investigator — Advanced Medical and Dental Institute, Universiti Sains Malaysia
Locations (1):
- Advanced Medical and Dental Institute (AMDI), Kepala Batas, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No